CLINICAL TRIAL: NCT00312598
Title: Investigation of Body Mass Index, Body Composition, Resting Energy Expenditure, Respiratory Quotient and Metabolic Changes Following a Switch From Olanzapine, Quetiapine or Risperidone to Aripiprazole
Brief Title: Body Mass Index (BMI) and Metabolic Changes Following Switch to Aripiprazole From Olanzapine, Risperidone and Quetiapine
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Karen Graham, MD, associate professor of psychiatry, University of North Carolina, Chapel Hill
Other Study IDs: IND 70,111; GCRC 2086
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Mood Disorders
Keywords: schizophrenia; BMI; weight; aripiprazole; antipsychotic; Mood Disorders with psychotic features
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mood Disorders; Body Weight | interventions — Aripiprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum collected at baseline and end of study to be assayed in the future for related metabolic tests which are not specified at this time.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- aripiprazole: observational measures of metabolic parameters of subjects who are making clinically determined medication switch to aripiprazole
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole
  Other Names: Abilify

SUMMARY:
Weight gain is a serious, common side effect of many antipsychotic medications. On average, the highest amounts of weight gain are found to occur in people taking clozaril and olanzapine, but with significant weight gain occuring in those on the other atypical antipsychotics as well.

We, the researchers at the University of North Carolina, propose an open-label observational, pilot study of the changes in weight, BMI, body composition, and lipids, glucose, insulin and other metabolic parameters occurring in subjects as they switch from treatment with olanzapine, risperidone or quetiapine to aripiprazole. This medication switch will be determined prior to their entering this study by their treating psychiatrist. We also will determine resting energy expenditure (REE) and respiratory quotient (RQ) as measured by metabolic cart to determine if either energy expenditure or the propensity to store energy as fat may be involved in any changes to weight that are detected. Food intake, hunger, and physical activity will also be assessed.

DETAILED DESCRIPTION:
Weight gain is a serious, common side effect of many antipsychotic medications. It is a frequent cause of poor adherence to antipsychotic medications and a major contributor to medical problems including Syndrome X, various cancers, osteoarthritis and sleep apnea. Syndrome X, also called the Metabolic Syndrome, is a constellation of abnormalities of metabolism that confer a high risk of coronary heart disease. Syndrome X includes glucose intolerance, dyslipidemia, hypertension, and central obesity. Long-term patients on antipsychotic medications have markedly increased rates of Syndrome X that are consistent with increased cardiovascular morbidity and decreased life expectancy.

A recent meta-analysis estimated weight gain at 10 weeks of treatment for a variety of antipsychotics and found that clozapine had the highest average weight gain (4.45 kg), followed by olanzapine (4.15 kg), quetiapine (2.2 kg), risperidone (2.18 kg), and ziprasidone (0.04 kg) . For some drugs weight gain continues over many months, with the time to plateau being directly related to the initial degree of weight gain. Early data for the most recently approved antipsychotic, aripiprazole, shows it to be weight neutral but the characteristics of its effects on weight are still to be determined. A recent publication of 224 subjects switching by three different switching strategies from haloperidol, thioridazine, risperidone or olanzapine to aripiprazole found weight loss of between 1.3 and 1.7 kg after 8 weeks on aripiprazole. Cholesterol levels improved in subjects switching from olanzapine to aripiprazole.

Atypical antipsychotic medications that can improve the factors associated with Syndrome X could offer a very attractive alternative for patients who have already developed this constellation of symptoms during treatment with other antipsychotics. It is not known if a switch to aripiprazole from an atypical antipsychotic medication that has caused excessive weight gain and/or abnormalities of glucose, lipids or blood pressure will result in significant improvement in these factors or simply halt worsening. If worsening is only halted, then switch from a weight-inducing drug to aripiprazole should be done early. If factors associated with Syndrome X can be reversed, then switch to aripiprazole would be very beneficial even after abnormalities have developed.

We propose an open-label pilot study of the changes in weight, BMI, body composition, and lipids, glucose, insulin and other metabolic parameters occurring in subjects as they switch from treatment with olanzapine, risperidone or quetiapine to aripiprazole. We also will determine resting energy expenditure (REE) and respiratory quotient (RQ) as measured by metabolic cart to determine if either energy expenditure or the propensity to store energy as fat may be involved in any changes to weight that are detected. Food intake, hunger, and physical activity will also be assessed.

Recruited subjects will enter a screening phase where patient eligibility is determined through assessments of psychiatric and physical health, including physical examination, blood tests and urine drug screen. Subjects not meeting eligibility criteria will be discontinued.

Thirty subjects will be enrolled into this open label study. At entry into the study, anthropometric measures (wt, ht, waist, hip), body composition, respiratory quotient (RQ), resting energy expenditure (REE), and measures of food intake, hunger, and physical activity will be assessed. Additionally, the Positive and Negative Symptom Scale (PANSS) will be used to assess clinical status and all women will have a blood pregnancy test as required prior to having a DXA scan. Following completion of these assessments, subjects will begin a two week cross-taper from their current antipsychotic to aripiprazole. Psychiatric symptoms, weight, medical status and medication query will be reassessed after 2, 4, 8 and 12 weeks. RQ and hunger will be reassessed at the 4 week time point. Fasting bloodwork, pregnancy test, urine drug screen, vital signs, and all baseline assessments will be repeated at the 12 week time point or at early termination. During the study, dosage of aripiprazole will be tailored to each subject's need based on symptoms and side effects, and will remain at or below the maximum recommended dosage.

ELIGIBILITY:
Inclusion Criteria:

* Any ethnicity
* Antipsychotic monotherapy with olanzapine, risperidone or quetiapine for minimum of 1 month at entry into study and with weight gain of 2 BMI units while on this medication or development of abnormalities of glucose (greater than 110 mg/dl fasting), lipids (total cholesterol [TC], high-density lipoprotein [HDL], triglycerides [TG], or low-density lipoprotein [LDL] greater than 10% change) or blood pressure (greater than 20 mmHg change in systolic or diastolic)
* Antipsychotic monotherapy with aripiprazole is planned by the subject's treating psychiatrist.
* Subjects able to fully participate in the informed consent process
* Female subjects of childbearing potential must be using a medically accepted means of contraception which includes tubal ligation, hysterectomy, condoms, oral contraceptives, intrauterine device (IUD), cervical cap, diaphragm, transdermal contraceptive patch, and abstinence.

Exclusion Criteria:

* Subjects have had a previous trial of aripiprazole
* Serious or unstable medical illness which requires ongoing treatment with medication. This does not include non-insulin dependent diabetes, dyslipidemia or hypertension.
* At serious suicidal risk.
* Subjects with substance abuse or dependence.
* Female subjects who are either pregnant or nursing.
* Known history of mental retardation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatry outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
BMI change | 12 weeks
Body composition change | 12 weeks
Change in laboratory markers of cardiovascular and diabetes risk | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Graham, MSc MD, Principal Investigator — University of North Carolina, Chapel Hill